CLINICAL TRIAL: NCT00253214
Title: Placebo-Controlled Evaluation of Galantamine in the Treatment of Alzheimer's Disease: Safety and Efficacy of a Controlled-Release Formulation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR006037
Record Dates: First submitted 2005-11-10; First posted 2005-11-15 (Estimated); Last update posted 2011-05-23 (Estimated); Status verified 2010-11

CONDITIONS: Alzheimer Disease; Dementia
Keywords: Alzheimer's disease; dementia; galantamine hydrobromide; controlled-release; once-daily dosing
MeSH Terms: conditions — Alzheimer Disease; Dementia | interventions — Galantamine

INTERVENTIONS:
Drug: galantamine hydrobromide

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness of a once daily controlled-release form of galantamine (a drug for treating dementia) versus placebo in the treatment of patients with Alzheimer's disease.

DETAILED DESCRIPTION:
Dementia is a chronic, progressive brain disease that may involve a number of symptoms, including memory loss and changes in personality, behavior, judgment, attention span, language and thought. The most common type of dementia is Alzheimer's disease. Over time, patients with Alzheimer's disease may lose the ability to perform daily tasks related to personal care (for example, bathing, dressing, and eating) and may be unable to handle money or travel to familiar places. Previous clinical trials have shown that a twice-daily dose of galantamine (18 - 32 mg/day) improved symptoms of Alzheimer's disease. This multicenter, double-blind, placebo-controlled study evaluates the safety and effectiveness of a controlled-release form of galantamine in patients with Alzheimer's disease. All patients receive placebo during the first month of the study. Patients then receive controlled-release galantamine (8 - 24 mg once daily), or immediate-release galantamine (4 - 12 mg twice daily) or placebo for 6 months. The dose of galantamine starts at 8 mg/day and may be increased up to 24 mg/day, if needed. The dose may be adjusted up or down during the first 12 weeks of double-blind treatment based upon effectiveness and tolerability. Patients continue to receive the dose they are taking at the end of 12 weeks for the remainder of the study. The primary measures of effectiveness include the change from baseline to the end of treatment in the ADAS-cog/11 (Alzheimer's Disease Assessment Scale: sum of 11 cognitive items) and CIBIC-plus (Clinician's Interview Based Impression of Change - Plus Caregiver Input) scores. Additional measures of effectiveness include the change from baseline in the Alzheimer's Disease Cooperative Study - Activities of Daily Living (ADCS-ADL) and the Neuropsychiatric Inventory (NPI) scores. Safety evaluations (incidence of adverse events, electrocardiograms (ECGs), physical examinations, laboratory tests) are performed throughout the study. Patients who complete the double-blind portion of the study have the opportunity to receive galantamine in an open-label follow-up study. Patients may also participate in an optional portion of the study in which their genetic material is analyzed to see if contains something that would affect the way galantamine is used by their bodies. The study hypothesis is that treatment with controlled-release galantamine is effective in improving the symptoms of Alzheimer's disease and is well tolerated. Controlled-release galantamine 8 - 24 mg by mouth once daily, or immediate-release galantamine 4 - 12 mg by mouth twice daily, or placebo. Dosing starts at 8 mg/day and may be increased up to 24 mg/day, if needed. The study duration is 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Outpatients with a diagnosis of mild-to-moderate Alzheimer's disease according to the National Institute of Neurological and Communicative Disorders and the Alzheimer's Disease and Related Disorders Association (NINCDS-ADRDA) criteria (including patients living in residential homes for the elderly or day patients)
* have a Mini-Mental Status Examination (MMSE) score of 10 - 24, and a score of at least 18 on the cognitive portion of the Alzheimer's Disease Assessment scale (ADAS-cog-11) with an onset between ages 40 and 90
* history of at least a 6 months of gradual and progressive cognitive decline
* have a consistent informant to accompany the patient on scheduled visits

Exclusion Criteria:

* Neurogenerative disorders such as Parkinson's disease
* cognitive impairment resulting from acute cerebral trauma, cerebral damage due to a lack of oxygen, vitamin deficiency, infections such as meningitis or AIDS, significant endocrine or metabolic disease, mental retardation or a brain tumor
* dementia caused by small strokes or cerebrovascular disease
* having epilepsy, significant psychiatric disease, active peptic ulcer, clinically significant liver, kidney or lung disorders, or heart disease
* females of child bearing potential without adequate contraception

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 973 (Actual)
Dates: Start 2001-03; Study Completion 2002-07 (Actual)

PRIMARY OUTCOMES:
Change from baseline to end of treatment for controlled release group in ADAS-cog/11 (Alzheimer's Disease Assessment Scale: sum of 11 cognitive items) and CIBIC-plus (Clinician's Interview Based Impression of Change - Plus Caregiver Input) scores

SECONDARY OUTCOMES:
Change from baseline in ADAS-cog/13, /10, /mem scores, NPI, and ADCS/ADL; safety and tolerability of controlled-release formulation; difference in effects between the controlled-release and immediate-release formulations

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.

REFERENCES:
- [Result] Brodaty H, Corey-Bloom J, Potocnik FC, Truyen L, Gold M, Damaraju CR. Galantamine prolonged-release formulation in the treatment of mild to moderate Alzheimer's disease. Dement Geriatr Cogn Disord. 2005;20(2-3):120-32. doi: 10.1159/000086613. Epub 2005 Jun 30. PMID 15990426
- [Derived] Lim AWY, Schneider L, Loy C. Galantamine for dementia due to Alzheimer's disease and mild cognitive impairment. Cochrane Database Syst Rev. 2024 Nov 5;11(11):CD001747. doi: 10.1002/14651858.CD001747.pub4. PMID 39498781
- See also: A study of the safety and effectiveness of a controlled-release form of galantamine in patients with Alzheimer's disease — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=703&filename=CR006037_CSR.pdf